CLINICAL TRIAL: NCT00683995
Title: A Phase III Clinical Study of KW-2246 for Breakthrough Pain in Cancer Patients
Brief Title: A Phase III Clinical Study of KW-2246
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2246-0703
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Pain, Cancer
Keywords: Pain, Cancer
MeSH Terms: conditions — Cancer Pain | interventions — Fentanyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): KW-2246 (fentanyl citrate)
  Interventions: Drug: KW-2246 (fentanyl citrate)

INTERVENTIONS:
Drug: KW-2246 (fentanyl citrate) — KW-2246 (fentanyl citrate)

SUMMARY:
This study is designed to assess the safety and efficacy of long-term KW-2246 treatment as rescue medication for breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in the study on a voluntary basis.
* Patients who have been eligible for the confirmatory trial by meeting the inclusion criteria applicable at the time of giving written informed consent and those applicable at the time of randomization, and who have completed the confirmatory trial.
* Outpatients who live with a caregiver such as a family member, or inpatients.
* Require rescue medication at least 0.5 times (at least once every two days) but not more than three times per day on average as determined by the investigator.
* Performance Status (ECOG) of 3 or less at the time of giving written informed consent.
* Have a life expectancy of at least three months as determined by the investigator.
* Be able to receive diary training and have been able to properly complete diaries during the confirmatory trial.

Exclusion Criteria:

* Have experienced intolerable adverse reactions (as defined in Attachment 3) during the confirmatory trial.
* Have met any of the exclusion criteria applicable at the time of giving written informed consent, those applicable at the time of randomization, or subject withdrawal criteria in the confirmatory trial.
* Serious respiratory dysfunction.
* Asthma.
* Serious bradyarrhythmia.
* Serious hepatic dysfunction.
* Serious renal dysfunction.
* Susceptibility to respiratory depression due to conditions such as increased intracranial pressure, head injury and brain tumor.
* Patients who have a history of clinically significant adverse reactions to the combination of opioid analgesics and any of the following drugs/substances, and who are currently receiving or expect to receive any of them during the study:

Central nervous system depressants (phenothiazines, benzodiazepines and barbiturates), inhalation anesthetics, monoamine oxidase inhibitors, tricyclic antidepressants, skeletal muscle relaxants, antihistamines, ritonavir, alcohol, itraconazole, amiodarone, clarithromycin, diltiazem, and fluvoxamine.

* History of convulsive seizures (except a single episode of infantile febrile convulsions).
* History of hypersensitivity to fentanyl.
* Pregnant or lactating women, possibly pregnant women, or women who are planning to become pregnant.
* Patients who are judged by the investigator/subinvestigator to be inappropriate for this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2008-03; Primary Completion 2009-07 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Kyowa Kirin Co., Ltd.
Locations (20):
- Japan (20):
  - Nagoya, Aichi-ken
  - Katori-shi, Chiba
  - Matsuyama, Ehime
  - Kitakyushu, Fukuoka
  - Kōriyama, Fukushima
  - Sapporo, Hokkaido
  - Nishinomiya, Hyōgo
  - Kasama, Ibaraki
  - Kanazawa, Ishikawa-ken
  - Uji, Kyoto
  - Azumino, Nagano
  - Ibaraki, Osaka
  - Izumisano, Osaka
  - Mibu, Tochigi
  - Bunkyo-ku, Tokyo
  - Shinagawa-ku, Tokyo
  - Kumamoto
  - Okayama
  - Toyama
  - Wakayama